CLINICAL TRIAL: NCT02642705
Title: New Treatment Modalities in Obese Patients: High Intensity Interval Training and Hypoxic Conditioning
Brief Title: High Intensity Interval Training and Hypoxic Conditioning in Obese Patients
Acronym: HYPINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A01482-45
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- High intensity interval training N (Experimental): High intensity interval training N: The intervention consists in 8-week exercise training, 3 times a week for one hour, according to a high intensity interval training protocol (1 min ON at 100% maximal power output, 1 min OFF), breathing ambient air (normoxia)
  Interventions: Other: High intensity interval training N
- High intensity interval training H (Experimental): High intensity interval training H: The intervention consists in 8-week exercise training, 3 times a week for one hour, according to a high intensity interval training protocol (1 min ON at 100% maximal power output, 1 min OFF), breathing hypoxic air (about 3 500 m of altitude)
  Interventions: Other: High intensity interval training H
- Constant load exercise training N (Active Comparator): Constant load exercise training N: The intervention consists in 8-week exercise training, 3 times a week for one hour, according to a constant load training protocol (50% maximal power output), breathing ambient air (normoxia)
  Interventions: Other: Constant load exercise training N
- Constant load exercise training H (Experimental): Constant load exercise training H: The intervention consists in 8-week exercise training, 3 times a week for one hour, according to a constant load training protocol (50% maximal power output), breathing hypoxic air (about 3 500 m of altitude)
  Interventions: Other: Constant load exercise training H
- Hypoxic conditioning at rest (Experimental): Hypoxic conditioning at rest : The intervention consists in 8-week conditioning period, 3 times a week, hypoxic breathing for one hour (about 4500 m of altitude) while seating quietly
  Interventions: Other: Hypoxic conditioning at rest
- Normoxic conditioning at rest (Sham Comparator): Normoxic conditioning at rest : The intervention consists in 8-week conditioning period, 3 times a week, normoxic breathing for one hour (ambient air) while seating quietly
  Interventions: Other: Normoxic conditioning at rest

INTERVENTIONS:
Other: High intensity interval training N — Exercise training and ambient air breathing
  Arms: High intensity interval training N
Other: High intensity interval training H — Exercise training and hypoxic breathing
  Arms: High intensity interval training H
Other: Constant load exercise training N — Exercise training and ambient air breathing
  Arms: Constant load exercise training N
Other: Constant load exercise training H — Exercise training and hypoxic breathing
  Arms: Constant load exercise training H
Other: Hypoxic conditioning at rest — Hypoxic breathing at rest
  Arms: Hypoxic conditioning at rest
Other: Normoxic conditioning at rest — Normoxic breathing at rest (placebo)
  Arms: Normoxic conditioning at rest

SUMMARY:
The present study aims at evaluating the effect of two innovative treatment strategies in obese patients: high intensity interval training and hypoxic conditioning. Obese patients will be randomized in groups performing high intensity interval training, constant load training, hypoxic conditioning or placebo normoxic conditioning for 8 weeks. The effects of the interventions will be measured regarding exercise tolerance, blood pressure, body composition, metabolic status.

DETAILED DESCRIPTION:
120 obese patients will be randomized to 6 intervention groups. Each group will follow an 8-week intervention (3 session per week) with either high intensity interval training in normoxia or hypoxia, constant load exercise training in normoxia or hypoxia, hypoxic or normoxic (placebo) conditioning at rest. Exercise capacity, metabolic status, blood pressure, vascular function and physical activity will be assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 35 kg/m²
* Physical activity <2 hours/week
* No chronic disease or treatment able to interfere with inflammation and metabolic perturbatiosn associated with obesity

Exclusion Criteria:

* Diabetes mellitus treated with insulin
* Auto-immune or inflammatory diseases requiring long term therapy
* Unstable dysthyroidism
* Bariatric surgery within the past 18 months
* Tumoral, inflammatory, infectious, cardiac, respiratory, kidney, digestive disease
* Untreated sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | 8 weeks
  Maximal oxygen consumption during an incremental exercise test

SECONDARY OUTCOMES:
Metabolic status | 8 weeks
  Blood lipids, glycemia, HOMA index, oxydative stress and inflammatory status
Body composition | 8 weeks
  MRI fat free mass and adipose tissue measurements
Blood pressure | 8 weeks
  24 h ambulatory blood pressure mesurement
Vascular function | 8 weeks
  Post-ischemic hyperemia (Endo-Pat) and pulse wave velocity
Physical activity | 8 weeks
  Spontaneous physical activity measured by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verges S, Chacaroun S, Godin-Ribuot D, Baillieul S. Hypoxic Conditioning as a New Therapeutic Modality. Front Pediatr. 2015 Jun 22;3:58. doi: 10.3389/fped.2015.00058. eCollection 2015. PMID 26157787
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531